CLINICAL TRIAL: NCT01325311
Title: Phase IIA, Randomized Placebo-Controlled Trial of Single High Dose Cholecalciferol and Daily Genistein (G-2535) Versus Placebo in Men With Early Stage Prostate Cancer Undergoing Prostatectomy
Brief Title: Cholecalciferol and Genistein Before Surgery in Treating Patients With Early Stage Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2013-00451; NCI-2013-00451 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UWI09-14-01; CDR0000698228; CO-10805; CO 10805 (Other: University of Wisconsin Hospital and Clinics); UWI09-14-01 (Other: DCP); N01CN35153 (NIH); P30CA014520 (NIH)
Record Dates: First submitted 2011-03-23; First posted 2011-03-29 (Estimated); Results first posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-06

CONDITIONS: Prostate Adenocarcinoma; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cholecalciferol; Genistein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (cholecalciferol, genistein) (Experimental): Patients receive cholecalciferol PO on day 1 and genistein PO QD on days 1-21 or 1-28. Patients then undergo prostatectomy.
  Interventions: Drug: Cholecalciferol; Drug: Genistein; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO on day 1 and placebo PO QD on days 1-21 or 1-28. Patients then undergo prostatectomy.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — Given PO
  Other Names: 9,10-Secocholesta-5,7,10(19)-trien-3-ol; Calciol; Delsterol; Vitamin D3
  Arms: Arm I (cholecalciferol, genistein)
Drug: Genistein — Given PO
  Other Names: 4',5, 7-Trihydroxyisoflavone; Genestein; Genisteol; Prunetol
  Arms: Arm I (cholecalciferol, genistein)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)

SUMMARY:
This randomized phase II trial studies cholecalciferol and genistein compared to placebo in treating patients with early stage prostate cancer. Cholecalciferol and genistein may slow the growth of cancer cells and may be an effective treatment for prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine differences in prostate tissue steady state concentrations of calcitriol in participants treated with a single dose cholecalciferol (200,000 IU) and G-2535 (which provides 600 mg of genistein) and those receiving placebo.

SECONDARY OBJECTIVES:

I. To determine the effect of each intervention arm and resulting prostate tissue levels of calcitriol on down-stream related biomarkers and related mechanistic pathways in blood and tissue.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive cholecalciferol orally (PO) on day 1 and genistein PO once daily (QD) on days 1-21 or 1-28. Patients then undergo prostatectomy.

ARM II: Patients receive placebo PO on day 1 and placebo PO QD on days 1-21 or 1-28. Patients then undergo prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have microscopic confirmation of adenocarcinoma of the prostate within three months of randomization; clinical stage T1 and T2 a, b, or c are allowed
* Participants' prostate cancer must be confined to the prostate (in the clinical judgment of the treating physician)
* Participants must be candidates for prostatectomy
* Participants must have Eastern Cooperative Oncology Group (ECOG) performance status =<1 (Karnofsky >= 70%)
* White blood cell (WBC) within normal limits
* Platelets >= 100 K/uL
* Hemoglobin >= 10 g/dL
* Thyroid-stimulating hormone (TSH) =< 4.20 uIU/mL
* Free T4 =< 12.5 ng/dL
* Bilirubin within upper limit of normal
* Aspartate aminotransferase (AST) =< 1.5 x upper limit of normal
* Creatinine =< 2.0 mg/dL
* Serum calcium: within institutional normal limits
* Participants must agree to stop taking nonsteroidal anti-inflammatory drugs (NSAIDS) during the course of the study, however, low dose aspirin (< 100 mg/day) will be allowed; no wash out period is required
* Participants must be willing to discontinue consuming soy products and ingesting vitamin supplements while participating in this study
* The effects of cholecalciferol and genistein on the developing human fetus at the recommended therapeutic doses are unknown; for this reason, participants must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation
* Participants must have the ability to understand and sign a consent form indicating the investigational nature of the treatment and its potential risks

Exclusion Criteria:

* Participants may not have received any prior therapy for prostate cancer including: chemotherapy, hormonal therapy, brachytherapy, or external radiation
* Participants may not be receiving concurrent systemic therapy for other cancers
* Participants may not be receiving any other investigational agents
* Participants may not be taking the following p450 inducers and inhibitors: carbamazepine, clarithromycin, fluconazole, fosphenytoin, itraconazole, ketoconazole, phenobarbital, phenytoin, rifabutin, rifampin
* Participants who took finasteride or dutasteride within 6 months of the pre-randomization biopsy, are currently taking finasteride or dutasteride, or are planning on taking these agents during study participation
* Participants with a history of allergic reactions attributed to genistein or placebo, or compounds of similar chemical or biologic composition
* Participants with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Participants requires thyroid replacement therapy; Note: participants with a history of thyroid disease > 5 years ago, with current normal thyroid function, will be considered eligible
* Participant has current, known nephrolithiasis or a history of nephrolithiasis within the past 5 years
* Participant has any history of sarcoidosis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Jarrard, Principal Investigator — University of Wisconsin, Madison
Locations (11):
- United States (11):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Minneapolis Veterans Medical Center, Minneapolis, Minnesota
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - University of Rochester, Rochester, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology San Antonio Research PA, San Antonio, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm II (Placebo) | Arm I (Cholecalciferol, Genistein)
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm II (Placebo) | Arm I (Cholecalciferol, Genistein) | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.75 (4.50) | 62.14 (4.26) | 61.40 (4.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Tissue Levels of Calcitriol Between the Placebo and Cholecalciferol/Genistein Arms
Description: This is a measure of calcitriol in prostate tissue comparing placebo and cholecalciferol/genistein
Time Frame: up to Day 35
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm II (Placebo) | Arm I (Cholecalciferol, Genistein)
Number analyzed (Participants) | 8 | 7
ng/mL | 0.045 (0.127) | 0.057 (0.150)
Statistical Analysis 1: Comparison: Arm II (Placebo) vs Arm I (Cholecalciferol, Genistein); Using the Student t-test. If the normality assumption is tenuous, an appropriate transformation of the data such as logarithm will be considered for Student t-test or a nonparametric test such as Wilcoxon rank-sum test will be used for comparison; Test type: Superiority or Other; p = 0.922, t-test, 2 sided

2. Secondary Outcome: Levels of Calcidiol in the Participants Serum
Description: This is measuring the amount of Calcidiol that was found in the participants blood Serum at baseline and end of study
Time Frame: Baseline and up to day 35
Population: Due to sample one participant in Arm 1 was not analyzed for this Outcome.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm II (Placebo) | Arm I (Cholecalciferol, Genistein)
Number analyzed (Participants) | 8 | 6
ng/mL
  Baseline | 20.5 (5.5) | 24.5 (9.3)
  Pre-Surgery | 19.2 (5.1) | 27.3 (10.0)

3. Primary Outcome: Detectability of Calcitriol Levels in Tissue Between the Placebo and Cholecalciferol/Genistein Arms
Description: To identify the amount of Calcitriol that is found in the tissue comparing Placebo and Cholecalciferol/Genistein
Time Frame: up to 35 days
Measure: Number; unit: participants
Arm/Group | Arm II (Placebo) | Arm I (Cholecalciferol, Genistein)
Number analyzed (Participants) | 8 | 7
participants
  Undetectable | 7 | 6
  Detectable | 1 | 1

4. Secondary Outcome: Levels of Calcitriol in Participants Serum
Description: This is measuring the amount of Calcitriol that was found in the participants blood Serum at baseline and end of study.
Time Frame: baseline and Up to Day 35
Population: Due to sample one participant in Arm 1 was not analyzed for this Outcome.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm II (Placebo) | Arm I (Cholecalciferol, Genistein)
Number analyzed (Participants) | 8 | 6
ng/mL
  Baseline | 0.5 (0.1) | 0.5 (0.2)
  Pre-Surgery | 0.5 (0.7) | 0.1 (0.4)

5. Secondary Outcome: PBMC CYP mRNA Expression of CYP24
Description: This is a measure of expression of CYP24 in comparing placebo to Cholecalciferol/genistein.
Time Frame: Baseline and Up to Day 35
Population: Due to sample two participant in Arm I and 2 participants in Arm II were not analyzed for this Outcome.
Measure: Geometric Mean (Standard Deviation); unit: Ratio to Baseline
Arm/Group | Arm II (Placebo) | Arm I (Cholecalciferol, Genistein)
Number analyzed (Participants) | 6 | 5
Ratio to Baseline | 3.054 (3.997) | 2.202 (4.071)

6. Secondary Outcome: PBMC CYP mRNA Expression of CYP27B1
Description: This is a measure of expression of CYP27B1 in comparing placebo to Cholecalciferol/genistein.
Time Frame: Up to Day 35
Measure: Geometric Mean (Standard Deviation); unit: Ratio to Baseline
Arm/Group | Arm II (Placebo) | Arm I (Cholecalciferol, Genistein)
Number analyzed (Participants) | 8 | 7
Ratio to Baseline | 1.656 (2.628) | 2.389 (3.511)

7. Secondary Outcome: Total PSA in Serum
Description: This is a measure of the concentration of PSA in the blood serum at baseline and at the end of study.
Time Frame: at Baseline and up to Day 35
Population: Due to sample one participant in Arm I was not analyzed for this Outcome.
Measure: Median (Standard Deviation); unit: ng/mL
Arm/Group | Arm II (Placebo) | Arm I (Cholecalciferol, Genistein)
Number analyzed (Participants) | 8 | 6
ng/mL
  Baseline | 8.7 (7.3) | 6.3 (1.7)
  Day 35 | 8.3 (6.7) | 5.8 (2.1)

8. Secondary Outcome: Serum Calcium Levels at Baseline and Pre-Surgery
Description: This is a measurement of calcium in the Blood serum at baseline and at the end of the study.
Time Frame: Baseline and Day 35
Population: Due to sample one participant in Arm I was not analyzed for this Outcome.
Measure: Mean (Standard Deviation); unit: ng/mL (absolute change)
Arm/Group | Arm II (Placebo) | Arm I (Cholecalciferol, Genistein)
Number analyzed (Participants) | 8 | 6
ng/mL (absolute change)
  Baseline | 10.5 (0.4) | 11.3 (1.8)
  Day 35 | 10.8 (0.9) | 10.9 (0.9)

9. Secondary Outcome: Total IGF-1 in Serum at Baseline and Pre-Surgery
Description: This is measuring the concentration of the Biomarker IGF-1 in blood serum at Baseline and at the end of the study.
Time Frame: Baseline and up to Day 35
Population: Due to sample one participant in Arm I was not analyzed for this Outcome.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm II (Placebo) | Arm I (Cholecalciferol, Genistein)
Number analyzed (Participants) | 8 | 6
ng/mL
  Baseline | 64.2 (11.5) | 66.3 (12.8)
  Day 35 | 60.6 (17.9) | 74.6 (14.0)

10. Secondary Outcome: Total IGF-2 in Serum at Baseline and Pre-Surgery
Description: This is measuring the concentration of the Biomarker IGF-2 in blood serum at Baseline and at the end of the study
Time Frame: Baseline and Up to Day 35
Population: Due to sample one participant in Arm 1 was not analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm II (Placebo) | Arm I (Cholecalciferol, Genistein)
Number analyzed (Participants) | 8 | 6
ng/mL
  Baseline | 770.4 (333.4) | 805.9 (193.5)
  Pre-Surgery | 605.0 (175.4) | 858.8 (112.7)

11. Secondary Outcome: Total IGFBP-3 in Serum at Baseline and Pre-Surgery
Description: This is measuring the concentration of the Biomarker IGFBP-3 in blood serum at Baseline and at the end of the study.
Time Frame: Baseline and Up to Day 35
Population: Due to sample one participant from Arm 1 was not analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm II (Placebo) | Arm I (Cholecalciferol, Genistein)
Number analyzed (Participants) | 8 | 6
ng/mL
  Baseline | 1838.9 (887.3) | 2004.5 (309.8)
  Day 35 | 1667.5 (788.9) | 1843.4 (443.3)

12. Secondary Outcome: Total PTH in Serum at Baseline and Pre-Surgery
Description: This is measuring the concentration of the Biomarker PTH in blood serum at Baseline and at the end of the study
Time Frame: Baseline and Up to Day 35
Population: Due to sample one participant in Arm I was not analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm II (Placebo) | Arm I (Cholecalciferol, Genistein)
Number analyzed (Participants) | 8 | 6
ng/mL
  Baseline | 143.4 (26.5) | 144.8 (37.8)
  Pre-Surgery | 151.1 (25.8) | 136.5 (72.9)

13. Secondary Outcome: Immunohistochemistry Measurements in Benign Prostate Tissue (BPT)
Description: The Immunohistochemistry measurement for: AR (Nucleus), VDR (Cytoplasm), p21 (Nucleus), PGE2 (Cytoplasm), TUNEL Pos (Nucleus), Caspase 3 (Cytoplasm), PSMA (Cytoplasm), IGF-1 and IGF-2 (Cytoplasm), Akt (Nucleus and Cytoplasm), and pAkt (nucleus and Cytoplasm)
  This is to serve as normalized control data to determine expression of protein.
  The normalized optical densities were measured as optical density per unit area by densitometric scanning using Vectra imaging system (Perkin Elmer).
  This Optical Density is based on fluorescence.
Time Frame: Up to Day 35
Measure: Mean (Standard Deviation); unit: Normalized Optical Density
Arm/Group | Arm II (Placebo) | Arm I (Cholecalciferol, Genistein)
Number analyzed (Participants) | 8 | 7
Normalized Optical Density
  AR (Nucleus) | -0.362 (0.294) | 0.414 (1.301)
  VDR (Cytoplasm) | -0.451 (0.410) | 0.515 (1.179)
  p21 (Nucleus) | -0.085 (1.070) | 0.097 (0.900)
  PGE2 (Cytoplasm) | -0.161 (1.023) | 0.184 (0.934)
  TUNEL Pos (Nucleus) | -0.168 (0.842) | 0.192 (1.122)
  Caspase 3 (Cytoplasm) | -0.308 (0.659) | 0.352 (1.178)
  PSMA (Cytoplasm) | 0.025 (1.231) | -0.029 (0.630)
  IGF-1 (Cytoplasm) | -0.295 (0.607) | 0.337 (1.220)
  IGF-2 (Cytoplasm) | -0.335 (0.763) | 0.383 (1.081)
  Akt (Nucleus) | -0.316 (0.618) | 0.361 (1.198)
  pAkt (Nucleus) | -0.114 (0.920) | 0.131 (1.068)
  Akt (Cytoplasm) | -0.249 (0.766) | 0.284 (1.142)
  pAkt (Cytoplasm) | -0.053 (1.004) | 0.061 (0.991)

14. Secondary Outcome: Immunohistochemistry Measurements in Prostate Cancer Tissue (PCA)
Description: The Immunohistochemistry measurement for: AR (Nucleus), VDR (Cytoplasm), p21 (Nucleus), PGE2 (Cytoplasm), TUNEL Pos (Nucleus), Caspase 3 (Cytoplasm), PSMA (Cytoplasm), IGF-1 and IGF-2 (Cytoplasm), Akt (Nucleus and Cytoplasm), and pAkt (nucleus and Cytoplasm)
  This is to serve as normalized case data to determine expression of protein.
  The normalized optical densities were measured as optical density per unit area by densitometric scanning using Vectra imaging system (Perkin Elmer).
  This Optical Density is based on fluorescence.
Time Frame: Up to day Day 35
Population: Due to sample in Arm II one participants data was not analyzed.
Measure: Mean (Standard Deviation); unit: Normalized Optical Density
Arm/Group | Arm II (Placebo) | Arm I (Cholecalciferol, Genistein)
Number analyzed (Participants) | 7 | 7
Normalized Optical Density
  AR (Nucleus) | -0.563 (0.481) | 0.563 (1.015)
  VDR (Cytoplasm) | -0.281 (0.657) | 0.281 (1.177)
  p21 (Nucleus) | -0.185 (0.489) | 0.185 (1.296)
  PGE2 (Cytoplasm) | -0.135 (0.969) | 0.135 (1.009)
  TUNEL Pos (Nucleus) | -0.363 (0.664) | 0.363 (1.119)
  Caspase 3 (Cytoplasm) | -0.103 (0.742) | 0.103 (1.194)
  PSMA (Cytoplasm) | -0.210 (0.966) | 0.210 (0.982)
  IGF-1 (Cytoplasm) | 0.155 (1.027) | -0.155 (0.943)
  IGF-2 (Cytoplasm) | 0.443 (1.102) | -0.443 (0.572)
  Akt (Nucleus) | -0.309 (0.903) | 0.309 (0.981)
  pAkt (Nucleus) | -0.291 (0.325) | 0.291 (1.302)
  Akt (Cytoplasm) | -0.379 (0.785) | 0.379 (1.024)
  pAkt (Cytoplasm) | -0.365 (0.377) | 0.365 (1.244)

15. Secondary Outcome: Percent of Participants With CYP24 and CYP27B1 SNPs (DNA From Paxgene)
Time Frame: up to Day 35
Measure: Number; unit: percentage of participants
Arm/Group | Arm II (Placebo) | Arm I (Cholecalciferol, Genistein)
Number analyzed (Participants) | 8 | 7
percentage of participants
  rs2209314- T/C | 37.5 | 42.86
  rs2209314- T/T | 62.5 | 57.14
  rs2248359- C/C | 37.5 | 42.86
  rs2248359- C/T | 37.5 | 57.14
  rs2248359- T/T | 25 | 0
  rs2296241- A/A | 37.5 | 14.29
  rs2296241- A/G | 35.5 | 71.43
  rs2296241- G/G | 25 | 14.29
  rs2762939- C/G | 37.5 | 28.57
  rs2762939- G/G | 62.5 | 71.43
  rs927650- C/C | 0 | 71.43
  rs927650- C/T | 50 | 14.29
  rs927650- T/T | 50 | 14.29
  rs703842- A/A | 50 | 14.29
  rs703842- A/G | 37.5 | 71.43
  rs703842- G/G | 12.5 | 14.29

ADVERSE EVENTS:
Arm/Group | Arm II (Placebo) | Arm I (Cholecalciferol, Genistein)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 4/8 | 5/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm II (Placebo) (N=8) | Arm I (Cholecalciferol, Genistein) (N=7)
hyperthyriodism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
fatigue (General disorders) | 1 (1) | 0 (0)
pain (General disorders) | 0 (0) | 1 (1)
sinusitis (Infections and infestations) | 0 (0) | 1 (2)
blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
increased serum chloride (Investigations) | 1 (1) | 0 (0)
platelet count decreased (Investigations) | 0 (0) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
sinus pain (Nervous system disorders) | 0 (0) | 1 (2)
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
calcified lung nodule-right ct scan (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less